CLINICAL TRIAL: NCT03435939
Title: Anti-Inflammatory Therapy to Augment CFTR Rescue in CF Patients
Brief Title: Effect of Losartan in Cystic Fibrosis (CF)-NIH Grant #133240
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Matthias Salathe, MD, Chairperson-Professor- Internal Medicine, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00146945
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- losartan (Experimental): a daily dose of 50 mg losartan for 7 days (for tolerability). Then, the losartan dose will be increased to 100 mg daily for 12 weeks.
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan — 50 mg/day for 7 days followed by 100 mg/day for 12 weeks
  Other Names: Cozaar

SUMMARY:
The goal of this study is to execute a small clinical proof of concept trial: To examine the effects of losartan on mucociliary clearance (MCC) in patients not eligible for CFTR rescue therapies

DETAILED DESCRIPTION:
CF is the most common inherited disease causing a shortened life span, affecting ~30,000 people in the United States with annual health care costs of at least $1.8 billion. The median age of predicted survival of these patients has improved and is now almost 40 years in the US. Over the last two decades, investigators have identified ~2,000 mutations in the CF transmembrane conductance regulator (CFTR) gene. These mutations are imperfectly classified into 5 groups, and small molecules are being developed that rescue group-specific CFTR mutants. These agents have produced remarkable improvements in some patients. The CFTR potentiator ivacaftor (Kalydeco™), approved by the FDA mainly for class III mutations especially G551D, improves ion transport (large decrease in sweat chloride), clinical outcome (increased FEV1 and weight, decreased exacerbations), and quality of life. Furthermore, the FDA recently approved Orkambi™ (a corrector and potentiator: lumacaftor plus ivacaftor) because it reduced exacerbation rates by up to 39% in patients homozygous for F508del.

It has been demonstrated in vitro that improvements in airway surface liquid (ASL) volume are highly predictive of changes seen in clinical studies and track with tracheal mucus velocities measured in sheep in vivo using the CFTR potentiator ivacaftor, inhaled hypertonic saline and other interventions (preliminary data). ASL volume is regulated by ion fluxes through ENaC, CFTR, CaCC, and BK channels, and TGF-β1-mediated inflammation in CF cells decreases activities of CaCC (8) and BK. These findings suggest that effective and safe anti-inflammatory therapy has the potential to improve mucociliary dysfunction in CF patients, even in the absence of small molecule therapy. Currently used anti-inflammatory therapies such as high-dose ibuprofen and steroids produce unwanted side effects that negate their effectiveness. Other medications showed severe side effects in clinical trials. However, experiments proposed in this application will test the hypothesis that losartan provides a safe and effective anti-inflammatory therapy needed to improve outcomes in CF patients.

Briefly, 16 patients with CF, >18 years of age, who are not on CFTR augmentation therapy will be recruited for this trial (4 per year). After signing informed consent at the screening visit, spirometry will be performed, take blood for safety and inflammatory markers, and test for pregnancy where applicable. Since losartan has teratogenic effects, strict birth control in female participants will be enforced. Eligible patients will complete visits as following:

Quality of life will be assessed by CF quality of life questionnaire - revised (CFQ-R). Cytokines will be measured from nasal fluid collected by Leukosorb filter paper. After assessing baselines, a daily dose of 50 mg losartan will be started, followed by a safety visit 7 days after treatment start (± 2 days). Then, the losartan dose will be increased to 100 mg daily until week 14. Since this trial assesses anti-inflammatory effects of 100 mg losartan, the total duration will be 14 weeks to achieve >12 weeks of treatment with losartan.

ELIGIBILITY:
Inclusion Criteria:

* CF patients with any known mutation combination not on CFTR augmentation therapy
* ≥18 years of age
* Severity of the Disease: Suitable patients will have mild to moderate lung disease, as defined by:

  * Pulmonary Function: Each patient must have an FEV1 ≥40% of predicted at the screening visit.
  * Hemoglobin saturation: Patients must have an oxygen saturation of >92% on room air as determined by pulse oximetry at the screening visit.
  * Produces sputum regularly (daily basis, at minimum)
* FEV1 ≥ 40% of predicted at screening visit
* Able to sign Informed consent
* Negative COVID-19 test within 72 hours prior to MCC testing

Exclusion Criteria:

* When enrolling female patients
* Not willing to adhere to strict birth control (combination of two methods)
* If female, patient must be non-pregnant and non-lactating, and those of childbearing potential must be using an acceptable method of birth control (i.e., an Intrauterine Contraceptive Device with a failure rate of <1%, hormonal contraceptives or a barrier method). If a female patient is abstinent, she must agree to use one of the acceptable methods if she becomes sexually active.
* Unstable lung disease: As defined by a change in medical regimen during the preceding 2 weeks or an FEV1 ≥15% below value within 3 months
* Received an investigational drug or therapy during the preceding 30 days
* Active or former smokers with less than 1 year since quitting, or >10 pack-year smoking history
* Unable to adequately complete study measures, including spirometry
* Intolerance to angiotensin receptor blockers (ARB)
* Treatment with angiotensin converting enzyme (ACE) inhibitor
* Regular use of NSAIDs or potassium supplementation, treatment with aliskiren, on anticoagulation
* Oral corticosteroid use within 6 weeks
* Exacerbation requiring treatment within 6 weeks
* Treatment of mycobacterial infections
* Significant hypoxemia (oxygen saturation <92% on room air and rest or use of continuous oxygen treatment), chronic respiratory failure by history (pCO2 > 45 mmHg), clinical evidence of cor pulmonale
* Untreated arterial hypertension (systolic blood pressure >140 mm Hg, diastolic blood pressure > 90 mmHg)
* Blood pressure less than 90 mm Hg systolic while standing
* Cardiac, renal (creatinine 1.5 times normal limit), hepatic (LFTs > 3x normal upper limit), neurological, psychiatric, endocrine or neoplastic diseases that are judged to interfere with participation in study
* Known renal artery stenosis
* Concomitant airway disorders other than CF, such as ABPA
* Subjects with prior thoracic surgery
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the PI, would make the subject inappropriate for enrollment.
* Patients using intermittent inhaled or oral antibiotics will be allowed to participate in this trial. Patients on chronic, cycling antibiotics will be required to have completed at least 2 full cycles of the prescribed antibiotic prior to enrollment and should be studied during the same phase of treatment (on or off) during each study period.
* Have had radiation exposure within the past year that would cause them to exceed Federal Regulations by participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Improvement of mucociliary clearance ( MCC) and cough clearance (CC) | 12 weeks treatment
  Losartan (100 mg for >12 weeks) will improve MCC+CC clearance in CF patients not on CFTR augmentation therapy in % of baseline

SECONDARY OUTCOMES:
Improvement on pulmonary function tests (in %predicted) | 12 weeks of treatment
  forced expiratory volume at one second (FEV1) in %predicted
Improvement on pulmonary function tests (in L) | 12 weeks of treatment
  forced expiratory volume at one second (FEV1) in liters
Decrease of inflammatory markers | 12 weeks
  Changes in serum inflammatory markers (hsCRP, WBC including absolute neutrophil count, %PMNs, serum amyloid A or SAA, calprotectin, GM-CSF, TGF-β active and total)
Nasal cytokine changes | 12 weeks
  Nasal cytokine changes (TGF-β1 active and total, TNF-α, IL-1β, IL-6, IL-8, IL-13, COX-2)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Salathe, MD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
since this study is a pilot study, participant data will not be shared to other researchers.